CLINICAL TRIAL: NCT03950453
Title: Preventing Childhood Obesity Through a Mindfulness-Based Parent Stress Intervention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2000023271; 1R01DK117651-01A1 (NIH)
Record Dates: First submitted 2019-04-22; First posted 2019-05-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Child Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: cohort study
Who Masked: Participant, Outcomes Assessor
Masking Description: participant and outcomes assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Parenting Mindfully for Health Nutrition (PMH) (Experimental): Parenting Mindfully for Health (PMH) + nutrition and physical activity counseling to promote healthy eating and physical activity in parent and child.
  Interventions: Behavioral: Parenting Mindfully for Health Nutrition (PMH)
- Contact Control Nutrition (C+N) (Active Comparator): Contact control intervention (C) + nutrition and physical activity counseling (N).
  Interventions: Behavioral: Contact Control Nutrition (C+N)
- Historical Control (WLC) non-randomized (Other): Non-randomized, historical control group with only assessments during intervention and follow-up period.
  Interventions: Other: Non-randomized historical control (WLC) assessment only

INTERVENTIONS:
Behavioral: Parenting Mindfully for Health Nutrition (PMH) — PMH will include included the following components:
  1. mindfulness strategies as outlined in the MBSR manual,
  2. mindful parenting concepts,
  3. mindful eating and awareness of family choices;
  4. self and child monitoring of food intake, PA and emotional reactivity;
  5. utilizing mindfulness for emotion regulation and distress tolerance,
  6. behavioral strategies of goal setting and implementing increasing frequency of healthy food intake and physical activity (PA)
  Arms: Parenting Mindfully for Health Nutrition (PMH)
Behavioral: Contact Control Nutrition (C+N) — Contact Control Group where parents engage in a quiet, relaxing, but stimulating activity and also nutrition counseling.
  Arms: Contact Control Nutrition (C+N)
Other: Non-randomized historical control (WLC) assessment only — Non-randomized, historical control group with only assessments during intervention and follow-up period.
  Other Names: assessment only group
  Arms: Historical Control (WLC) non-randomized

SUMMARY:
This study will examine the mediator/moderator variables that affect efficacy of a parent stress intervention with nutrition education (PMH+N: parenting mindfully for health) vs. Control intervention with nutrition education (CTL+N) on parent stress, parenting, health behaviors and child obesity risk. A non-randomized historical control group will also be assessed during the intervention and follow-up periods throughout to obtain outcome assessment without any interventions being provided.

DETAILED DESCRIPTION:
This is a 5-year interdisciplinary project to assess a 12-week Parenting Mindfully for Health (PMH) + nutrition counseling (N) versus contact control intervention (C) + nutrition counseling (N), to examine short-term and long term enduring effects of PMH+N to promote healthy eating and physical activity in parent and child, and prevent childhood obesity risk in 2-5 year olds, via changes in parent stress and parenting. A non-randomized historical control group will also be assessed during the intervention and follow-up periods throughout to obtain outcome assessment without any interventions being provided.

ELIGIBILITY:
Inclusion Criteria:

* Family with a child between 2-5 years
* BMI of parent ≥30kg/m2
* Parents aged 18 yrs or older
* High parent stress (PSS mean score ≥25)
* Low income family as determined by HHS Poverty Guidelines

Exclusion Criteria:

* Diagnosis of mental retardation, autism or other pervasive developmental disorder for child;
* Current serious psychiatric or medical disorder requiring immediate treatment, including active alcohol or substance use disorders (confirmed by urine toxicology screening and history), psychotic illnesses, suicidal ideation, untreated diabetes, cardiovascular disease, cancers or any other active current illnesses that preclude study participation for child or parent;
* Inadequate English proficiency to complete questionnaires.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 246 (Actual)
Dates: Start 2018-11-11 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Parent Stress change from Pre to Post intervention | Baseline Pre-intervention to Post intervention at 12 weeks
  Parent stress measured by the Perceived Stress Scale scores ranging from 0-56 with higher scores indicating more stress.
Child BMI change post intervention and at short term 6 month follow-up | Change from Pre-intervention to post-intervention (week 12) and at 6 month short term follow up
  Child height will be measured with a measuring tape. For children, weight and height will be plotted on the CDC growth chart for the child's age to determine the BMI-for-age percentile scores.
Child food intake change | Baseline Pre-intervention and at post-intervention (week 12)
  Parent report of child food frequency questionnaire assessment of frequency of healthy and unhealthy food intake.
Parenting Behavior Change | TWT parenting behavior ratings at Baseline Pre-intervention and at post-intervention (week 12)
  Observed parenting behavior ratings for increase in positive parenting behaviors in the Toy Wait Task (TWT)

SECONDARY OUTCOMES:
Parent Stress change from Post intervention to follow up period over 24-months | Post intervention at 12 weeks to follow-up timepoints at 6-, 12-, 18- and 24- month timepoints
  Parent stress measured by the Perceived Stress Scale scores ranging from 0-56 with higher scores indicating more stress.
Child BMI change at long term term follow-up | Baseline compared to 12-month, 18-month and 24-month timepoint
  Child height will be measured with a measuring tape. For children, weight and height will be plotted on the CDC growth chart for the child's age to determine the BMI-for-age percentile scores.
Child food intake change | Baseline Pre-intervention and at post-intervention (week 12)
  Parent report of child food frequency questionnaire assessment of frequency of healthy and unhealthy food intake.
Parenting Stress Inventory (PSI) | PSI scores at Baseline Pre-intervention and at post-intervention (week 12) and at follow-ups months 6-, 12-, 18- and 24 month timepoints
  Parent reported PSI scores ranging from 18-90 with higher scores indicating higher parenting stress.

OTHER OUTCOMES:
Parent BMI | baseline
  Parent height will be measured with a stadiometer, and parent BMI will be calculated from weight and height. For parents, waist circumference (WC) and percent body fat will also be measured using the TANITA and following the well-established NHBLI and NHANES III protocol.
Parent BMI | at 12 week timepoint
  Parent height will be measured with a stadiometer and parent BMI will be calculated from weight and height. For parents, waist circumference (WC) and percent body fat will also be measured using the TANITA and following the well-established NHBLI and NHANES III protocol.
Parent BMI | at 6 month timepoint
  Parent height will be measured with a stadiometer and parent BMI will be calculated from weight and height. For parents, waist circumference (WC) and percent body fat will also be measured using the TANITA and following the well-established NHBLI and NHANES III protocol.
Parent BMI | at 12 month timepoint
  Parent height will be measured with a stadiometer and parent BMI will be calculated from weight and height. For parents, waist circumference (WC) and percent body fat will also be measured using the TANITA and following the well-established NHBLI and NHANES III protocol.
Parent BMI | at 18 month timepoint
  Parent height will be measured with a stadiometer and parent BMI will be calculated from weight and height. For parents, waist circumference (WC) and percent body fat will also be measured using the TANITA and following the well-established NHBLI and NHANES III protocol.
Parent BMI | at 24 month timepoint
  Parent height will be measured with a stadiometer and parent BMI will be calculated from weight and height. For parents, waist circumference (WC) and percent body fat will also be measured using the TANITA and following the well-established NHBLI and NHANES III protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Rajita Sinha, Principal Investigator — Yale University
Locations (1):
- The Yale Stress Center: Yale University, New Haven, Connecticut, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-07-05): https://cdn.clinicaltrials.gov/large-docs/53/NCT03950453/ICF_000.pdf